CLINICAL TRIAL: NCT07012759
Title: Novel Pleural Effusion Biomarkers Screening and Evaluation in Lung Adenocarcinoma Patients
Brief Title: Pleural Effusion Biomarkers in Lung Adenocarcinoma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Assistant Professor, Fu Jen Catholic University
Other Study IDs: FJUH113386
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Biomarkers; Lung Adenocarcinoma; Pleural Effusion
Keywords: Pleural effusion; biomarkers; lung cancer; clinical diagnosis
MeSH Terms: conditions — Adenocarcinoma of Lung; Pleural Effusion; Lung Neoplasms | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients with pleural effusion diagnosed as lung adenocarcinoma.
  Interventions: Other: biomarkers
- Control group: Patients with pleural effusion diagnosed as non-malignant.
  Interventions: Other: biomarkers

INTERVENTIONS:
Other: biomarkers — pleural effusion biomarkers in lung adenocarcinoma

SUMMARY:
This project aims to assess the expression levels of novel molecular markers identified through screening in clinical samples of malignant pleural effusion, to evaluate the feasibility and clinical utility of these markers as potential diagnostic genes for lung adenocarcinoma.

DETAILED DESCRIPTION:
Background： Pleural effusion is characterized by abnormal fluid accumulation within the pleural cavity. Patients with pleural effusion commonly present with symptoms such as thoracic tightness, dyspnea, cough, and thoracic pain. The etiology of pleural effusion is multifactorial, encompassing conditions such as tuberculosis infection, heart failure, autoimmune disorders, and malignancies. When cancer cells invade the pleural space, malignant pleural effusion occurs. Common primary sites of pleural effusion include the lungs, breasts, ovaries, and gastrointestinal tract. Hence, precise diagnosis and etiological determination are imperative for guiding therapeutic interventions and optimizing patient outcomes. Although the diagnosis of malignant pleural effusion predominantly relies on biomarkers, there remains scope for enhancing the sensitivity and specificity of traditional biomarkers.

Study Design： This study is a two-year, single-center, prospective case-control research Methods： The study plans to collect 100 cases of malignant and non-malignant pleural effusion samples from clinical patients. The molecular marker analysis will be performed on the supernatant and sedimented cells obtained through centrifugation. The investigator will compare the expression levels of marker genes previously identified in lung cancer cell models between malignant and non-malignant pleural effusion samples. The concentration of secretory proteins in the supernatant of pleural effusion will be analyzed using immunoblot assay, and the intracellular proteins will be analyzed using immunohistochemical staining.

Effect： Based on the experimental results, The investigator aim to identify novel diagnostic molecules for malignant pleural effusion and combine them with other diagnostic markers to enhance the sensitivity and specificity of clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring thoracentesis for pleural effusion drainage as determined by a physician based on clinical need.
* Signed informed consent.

Exclusion Criteria:

* Patients under the age of 18.
* Patients with malignancies other than lung adenocarcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The control group consists of non-malignant pleural effusion, while the case group includes those diagnosed with pleural effusion with lung adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
target gene expression levels between malignant and non-malignant pleural effusions | 20 minutes
  Novel biomarkers specifically expressed in malignant pleural effusions may provide additional diagnostic options for malignant lung cancer in clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No